CLINICAL TRIAL: NCT07231419
Title: A Phase 3, Randomized, Double-blind, Placebo-Controlled Study of the Efficacy and Safety of Suzetrigine in Subjects With Pain Associated With Diabetic Peripheral Neuropathy
Brief Title: Evaluation of Efficacy and Safety of Suzetrigine (SUZ) for Pain Associated With Diabetic Peripheral Neuropathy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX24-548-111
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Peripheral Neuropathic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Suzetrigine (SUZ) (Experimental): Participants will be randomized to receive SUZ.
  Interventions: Drug: Suzetrigine
- Placebo (Placebo Comparator): Participants will be randomized to receive placebo matched to SUZ.
  Interventions: Drug: Placebo (matched to SUZ)

INTERVENTIONS:
Drug: Suzetrigine — Tablets for oral administration
  Other Names: VX-548; SUZ
  Arms: Suzetrigine (SUZ)
Drug: Placebo (matched to SUZ) — Placebo matched to SUZ for oral administration.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of Suzetrigine in participants with pain associated with diabetic peripheral neuropathy (DPN).

ELIGIBILITY:
Key Inclusion Criteria:

* Body weight greater than or equal to (≥)45 kilogram (kg)
* Body mass index (BMI) ≥18 to less than (<) 40 kilogram per meter square (kg/m^2)
* Diagnosis of diabetes mellitus type 1 or type 2 and with glycosylated hemoglobin A1c (HbA1c) ≤9% and the presence of bilateral pain in lower extremities due to DPN for at least 1 year
* Weekly average of daily NPRS score ≥4 and less than or equal to (≤) 9 with limited variation in the 7-day Baseline Period

Key Exclusion Criteria:

* More than 3 missing daily NPRS scores during the 7-day Baseline Period
* Received Journavx within 30 days of study drug dosing
* Any sensory abnormality (excluding DPN) as pre-specified in the protocol

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 734 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2027-04-06 (Estimated); Study Completion 2027-04-06 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the Weekly Average of Daily Pain Intensity on the Numeric Pain Rating Scale (NPRS) at Week 12 Compared to Placebo | From Baseline up to Week 12

SECONDARY OUTCOMES:
Change From Baseline in the Medical Outcomes Study 36-item Short-form Health Status (SF-36v2) Physical Component Summary (PCS) Score at Week 12 Compared to Placebo (Pooled with data from Study VX24-548-110) | From Baseline up to Week 12

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Long Beach Research Institute, Long Beach, California
  - Velocity Clinical Research -San Bernardino, San Bernardino, California
  - Paradigm Clinical Research - Wheat Ridge, Wheat Ridge, Colorado
  - Velocity Clinical Research - Washington DC, Washington D.C., District of Columbia
  - Accel Research - Deland, DeLand, Florida
  - Velocity Clinical Research - Hallandale Beach, Hallandale, Florida
  - CNS Healthcare - Jacksonville, Jacksonville, Florida
  - Health Awareness, Inc. - Jupiter, Jupiter, Florida
  - 3Sync Research -Miami Lakes, Miami Lakes, Florida
  - Accel Research - Decatur, Decatur, Georgia
  - Healthcare Research Network - Flossmoor IL, Tinley Park, Illinois
  - Healthcare Research Network - Hazelwood MO, Hazelwood, Missouri
  - AMR Kansas City, Kansas City, Missouri
  - Brooklyn Clinical Research, Brooklyn, New York
  - Velocity Clinical Research - Syracuse, East Syracuse, New York
  - West Clinical Research, Morehead City, North Carolina
  - Velocity Clinical Research - Cleveland, Beachwood, Ohio
  - Velocity Clinical Research - Medford, Medford, Oregon
  - Velocity Clinical Research - Providence, East Greenwich, Rhode Island
  - Velocity Clinical Research - Spartanburg, Spartanburg, South Carolina
  - Zenos Clinical Research, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/